CLINICAL TRIAL: NCT03647345
Title: Investigation for Individualized Noninvasive Neuromodulation in Mild Cognitive Impairment
Brief Title: Noninvasive Dual-mode Stimulation Therapy for Neurorehabilitation in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-01-132-005
Record Dates: First submitted 2018-01-03; First posted 2018-08-27 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Noninvasive brain stimulation; Repetitive Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1: Anodal Dual-mode stimulation (Experimental): 10Hz of rTMS was applied over the left DLPFC for 10 minutes with simultaneous application of anodal tDCS on the right DLPFC.
  Each participant's 2-back verbal/nonverbal working memory task and variety cognitive function test are assessed and their resting-state fMRI data at three times: prior to stimulation (pre-stimulation), immediately after stimulation (post-stimulation) and 2 months after stimulation (f/u) are acquired.
  Interventions: Device: High-frequency rTMS on left DLPFC+anodal tDCS on right DLPFC
- Experimental 2: Cathodal Dual-mode stimulation (Experimental): 10Hz of rTMS was applied over the left DLPFC for 10 minutes with simultaneous application of cathodal tDCS on the right DLPFC.
  Each participant's 2-back verbal/nonverbal working memory task and variety cognitive function test are assessed and their resting-state fMRI data at three times: prior to stimulation (pre-stimulation), immediately after stimulation (post-stimulation) and 2 months after stimulation (f/u) are acquired.
  Interventions: Device: High-frequency rTMS on left DLPFC+cathodal tDCS on right DLPFC
- Active Comparator: Single sham stimulation (Active Comparator): 10Hz of rTMS was applied over the left DLPFC for 10 minutes with simultaneous application of tDCS with sham mode (no stimulation) on the right DLPFC.
  Each participant's 2-back verbal/nonverbal working memory task and variety cognitive function test are assessed and their resting-state fMRI data at three times: prior to stimulation (pre-stimulation), immediately after stimulation (post-stimulation) and 2 months after stimulation (f/u) are acquired.
  Interventions: Device: High-frequency rTMS on left DLPFC+sham tDCS on right DLPFC

INTERVENTIONS:
Device: High-frequency rTMS on left DLPFC+anodal tDCS on right DLPFC — 10Hz rTMS over the left DLPFC and anodal tDCS over the right DLPFC are simultaneously stimulated.
  Arms: Experimental 1: Anodal Dual-mode stimulation
Device: High-frequency rTMS on left DLPFC+cathodal tDCS on right DLPFC — 10Hz rTMS over the left DLPFC and cathodal tDCS over the right DLPFC are simultaneously stimulated.
  Arms: Experimental 2: Cathodal Dual-mode stimulation
Device: High-frequency rTMS on left DLPFC+sham tDCS on right DLPFC — 10Hz rTMS over the left DLPFC and sham tDCS (no stimulation) over the right DLPFC are simultaneously stimulated.
  Arms: Active Comparator: Single sham stimulation

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) or transcranial direct current stimulation (tDCS) has been used for the modulation of mild cognitive impairment (MCI) patients' cognitive function by altering the cortical excitability. Recently, more challenging approaches, such as stimulation of two or more sites or use of dual modality have been studied in MCI patients. In this study, simultaneous stimulation using both facilitatory rTMS (10Hz) and anodal or cathodal tDCS (dual-mode stimulation) over bilateral dorsolateral prefrontal cortices (DLPFCs) was investigated to compare its modulatory effects with single facilitatory rTMS stimulation in mild cognitive impairment patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild cognitive impairment diagnosed via a history, a neurocognitive test, and brain imaging

Exclusion Criteria:

* K-MMSE score under 9
* Major active neurological disease or psychiatric disease
* A history of seizure
* Metallic implants in their brain

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04-26 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of 2-back verbal working memory task | Change from Pre-intervention at 2 months
  Accuracy (percentile) of 2-back verbal working memory task

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No